CLINICAL TRIAL: NCT06839157
Title: An Artificial Intelligence - Assisted Model for Predicting Optimal Timing of Surgery in Advanced Ovarian Cancer: the Combined Study of the SUNNY Trial and the Real World Data
Brief Title: Artificial Intelligence - Assisted Model for Optimal Timing of Surgery in Advanced Ovarian Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai Gynecologic Oncology Group (Other Government)
Collaborators: Shanghai Zhongshan Hospital (Other); Cancer Hospital of the University of Chinese Academy of Sciences (Zhejiang Cancer Hospital) (Unknown); Sun Yat-sen University Cancer Centre (Unknown); Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: SUNNY-AI
Record Dates: First submitted 2025-02-18; First posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Ovarian, Fallopian, and Primary Peritoneal Cancer; Artificial Intelligence (AI)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cohort 1- SUNNY RCT Trial: 489 patients who were enrolled and randomized in the SUNNY RCT trials.
- Cohort 2- Pragmatic Trial: 4000 patients who were newly diagnosed as stage IIIC or IV primary epithelial ovarian cancer, fallopian tube cancer, or primary peritoneal cancer between 2015 and 2024

SUMMARY:
This study integrates data from the randomized controlled SUNNY trial (RCT) and real-world (RWD) data, and employs multimodal data fitting to construct a medical artificial intelligence model to identify the clinical characteristics of patient subgroups suitable for primary debulking surgery (PDS) or interval debulking surgery (IDS), and the cutoff values for selecting different timings of surgery for advanced ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients who were included in the SUNNY study or who were newly diagnosed with stage IIIC or IV primary epithelial ovarian cancer, fallopian tube cancer, or primary peritoneal cancer during the SUNNY study period (2015-2023)
* Underwent primary debulking surgery or interval debulking surgery
* Data avaliable on first-line treatment and follow-up

Exclusion Criteria:

* Non-epithelial ovarian cancer or borderline tumors.
* Low-grade tumors.
* Mucinous ovarian cancer.
* Missing data on first-line treatment and follow-up

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were included in the SUNNY study or who were newly diagnosed with stage IIIC or IV primary epithelial ovarian cancer, fallopian tube cancer, or primary peritoneal cancer during the SUNNY study period (2015-2023)
Sampling Method: Non-Probability Sample
Enrollment: 4489 (Estimated)
Dates: Start 2027-03 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
The accuracy of predicting the 3-year overall survival (OS) difference between primary debulking surgery (PDS) and interval debulking surgery (IDS). | 3 years